CLINICAL TRIAL: NCT05371548
Title: Evaluating the Effectiveness of the Smart About Meds (SAM) Medication Management Mobile Application: A Randomized Controlled Trial
Brief Title: Smart About Meds (SAM) RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robyn Tamblyn (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Robyn Tamblyn, Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-7858
Record Dates: First submitted 2022-04-25; First posted 2022-05-12 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Medication Adherence
Keywords: medication adherence; mobile application; medication management; patient empowerment; randomized controlled trial
MeSH Terms: conditions — Medication Adherence; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (SAM app) (Experimental): Patients will receive training in and access to the SAM app at discharge. SAM uses prescribed and dispensed medication data to display a continuously updated drug list and provides patients and caregivers with tools to address barriers to adherence.
  Drug information: Provides patient-friendly drug monographs. Interaction checker: Generates drug-drug interactions between the patient's medications and other OTC drugs.
  Adherence alerts: Uses decision algorithms to alert users to adherence problems with the new regimen.
  Side effect checker: Displays possible side effects for each medication and frequency of occurrence.
  PIMs alerts: Alerts patients to potentially inappropriate medications in their list.
  Pharmacist connect: Connects users with pharmacists through a secured messaging service.
  Social connect: Allows users to share medication experiences. Caregiver connect: Allows patients to enroll caregivers who can use the app. Weekly medication schedule & pill reminders
  Interventions: Device: SAM mobile application
- Control (usual care) (No Intervention): Patients will receive usual care at discharge. On study units, medication reconciliation is conducted for all patients. Patients have their community medication list obtained via fax from their community pharmacy. The list is validated by the unit pharmacist who then reconciles it with admission orders, and recommends changes as needed to the attending physician. At discharge, the community drug list is reconciled with medications administered in hospital and the discharge prescription is generated by the attending physician or resident, classifying each medication as new medication, dose modification, discontinued therapy, or continued community medication. The discharge prescription is provided to the patient. Patients fill their discharge prescription at their community pharmacy. If there are questions about changes to the community drug list, the pharmacist will ask the patient, and if not clear will contact the discharging physician.

INTERVENTIONS:
Device: SAM mobile application — See description of intervention group
  Arms: Intervention (SAM app)

SUMMARY:
Introduction:

Almost half of patients discharged from hospital are re-admitted or return to the emergency department (ED) within 90 days. Patient nonadherence to medication changes during hospitalization and the use of potentially inappropriate medications (PIMs) both contribute to the risk of adverse events post-discharge. Smart About Meds (SAM) is a patient-centered mobile application designed to target medication nonadherence and PIMs use. This protocol describes a randomized controlled trial (RCT) to evaluate the effectiveness of SAM.

Methods & Analysis:

A pragmatic, stratified RCT will be conducted among 3,250 patients discharged from internal medicine, cardiac care, cardiac surgery, vascular surgery, and respiratory units of the Royal Victoria Hospital and the Montreal General Hospital. At discharge, patients will be randomized 1:1 to usual care or the SAM intervention. SAM integrates novel user-centered features (e.g. continuously updated medication list with pill images, side-effect checker, interaction checker) with pharmacist monitoring to tackle post-discharge nonadherence to new medication regimens. SAM also notifies patients of PIMS in their regimen, with advice to discuss with their physician.

Following discharge, patients will be followed for 90 days, during which the occurrence of the composite outcome of ED visits, hospital readmissions, or death will be measured. Secondary outcomes will include the individual components of the composite outcome, nonadherence to medication changes, defined as failure to fill a new prescription, filling a modified prescription at the incorrect dose, or filling discontinued medications, secondary medication adherence, patient empowerment, and health-related quality of life.

An intention-to-treat analysis will evaluate the effectiveness of SAM. Multivariable logistic regression will estimate differences between treatment groups in the proportion of patients nonadherent to at least one medication change. With a sample size of 3,250, there will be 80% power to detect a 5% absolute reduction in this outcome. Two-way interaction terms will test hypothesized modifiers of SAM's effectiveness, including hospital, unit, age, sex, gender and comorbidity burden. Binary and continuous secondary outcomes will be assessed using multivariable logistic and linear regression, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Covered by provincial (RAMQ) health insurance plan
* Covered by provincial (RAMQ) prescription drug insurance plan
* Owns a smartphone or tablet with internet connection
* At least one medication prescribed at discharge
* Speak and read English or French
* Age 18+

Exclusion Criteria:

* Discharged to rehabilitation center or to long-term care
* Transferred to a non-study unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3250 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
ED visits, hospital readmissions, and deaths (composite) | 90 days post-discharge
  This is a composite, binary outcome of having experienced an ED visit, hospital readmission, or death in the 90 days post-discharge. In Quebec, physicians must record the location of the services they provide to be remunerated on a fee-for-service basis. These medical services claims data are timely and accurate in measuring hospitalization occurrence and length of stay. The hospitalization database, which records admission and discharge diagnoses and procedures for all acute care hospitalizations in Quebec, will be used to collect additional descriptive information on the reasons for hospitalization and to re-validate the medical services data. Patients will be classified as having an ED visit or hospital readmission if they received a service whose location is recorded as an ED or inpatient hospital unit, respectively. Post-discharge deaths will be retrieved from the RAMQ beneficiary database.

SECONDARY OUTCOMES:
Individual components of the primary composite outcome | 90 days post-discharge
  ED visits, hospital readmissions and deaths occurring in the 90 days post-discharge, each of which will be measured separately as a binary secondary outcome.
Nonadherence to medication changes | 90 days post-discharge
  This is a binary outcome of a patient having adhered or not to medication changes in the discharge prescription. Nonadherence to medication changes is defined as a failure to fill a new prescription within 90 days of discharge, filling a modified prescription at the incorrect dose, or filling any discontinued medication in 90 days.
Secondary adherence | 90 days post-discharge
  Disease-modifying medications are defined as those that prevent health deterioration and typically need to be taken on a daily basis to be effective. A list of these medications will be compiled based on the World Health Organization's list of essential medicines. Secondary adherence will be measured for each disease-modifying medication that is filled using the medication possession ratio, which is calculated as the days of supply (based on the duration of dispensed prescription during follow-up) divided by the number of days of follow-up. Left-over supply prior to admission, when relevant, will be included in the calculation and only supply within the 90-day period for post-discharge dispensations will be included. In Quebec, over 94% of prescriptions are dispensed for 30 days or less, which should provide an accurate measure of persistence.
Patient and caregiver empowerment | 90 days post-discharge
  Patient and caregiver empowerment will be measured using the Patient Reported Outcome Measurement Information System (PROMIS) Self-Efficacy Measure for Managing Medication and Treatments (PROMIS-SE Meds). This 8-item measure assesses patient confidence in managing medication schedules of varying complexity and in challenging situations, such as when running out of supply or when adverse effects occur. Five-point ratings scales assess confidence levels. Scores are calibrated as T-scores (mean 50, SD 10), where higher scores indicate greater self efficacy.
Patient health-related quality of life | 90 days post-discharge
  Patient health-related quality of life (HRQoL) will be measured using the Patient Reported Outcome Measurement Information System-29 (PROMIS-29), which measures quality of life in seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance). Five-point ratings scales assess HRQoL. Scores are calibrated as T-scores (mean 50, SD 10), where higher scores indicate greater self HRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Researchers can request access to a trial dataset by contacting the PI or Research Project Manager. The dataset will include de-identified, processed participant data that underly the results reported in the main trial publication. Requesting researchers must ensure that their proposed use of the data has been approved by an independent review committee. A Data Transfer Agreement will govern the transfer of the data, the use of the data by the recipient, and the rights and obligations of both parties.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of the main trial results.
URL: https://mchi.mcgill.ca/

REFERENCES:
- [Derived] Tamblyn R, Habib B, Buckeridge DL, Weir DL, Frolova E, Alattar R, Rogozinsky J, Beauchamp C, Pupo R, Bartlett SJ, McDonald E. Evaluating the effectiveness of the Smart About Meds (SAM) mobile application among patients discharged from hospital: protocol of a randomised controlled trial. BMJ Open. 2024 Nov 24;14(11):e084492. doi: 10.1136/bmjopen-2024-084492. PMID 39581737